CLINICAL TRIAL: NCT06585397
Title: ICF-Based Evaluation of the Upper Extremity in Children With Quadriparetic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Neslihan Yildizdagi, Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: Neslihan Yildizdagi
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Upper Extremity Spasticity; Quadriplegic Cerebral Palsy
Keywords: ICF; Body structure and function; Activity; participation; cerebral palsy; upper extremity
MeSH Terms: conditions — Motor Activity; Cerebral Palsy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upper extremity evaluation of children with quadriparetic CP: Within the framework of ICF, the Modified Ashworth Scale, the Manual Ability Classification System and the Functional Independence Measure for Children will be applied to 20 quadriparetic children with CP.
  Interventions: Other: Grup 1

INTERVENTIONS:
Other: Grup 1 — Within the framework of ICF, the Modified Ashworth Scale, the Manual Ability Classification System and the Functional Independence Measure for Children will be applied to 20 quadriparetic children with CP.

SUMMARY:
Cerebral palsy (CP) is a neurodevelopmental disorder characterized by abnormalities in muscle tone, movement, and motor skills resulting from permanent, non-progressive damage to the developing brain before, during, or after birth. The worldwide prevalence of CP is 2-3 per 1000 live births. Spastic CP accounts for approximately 85% of all CP cases. Among the types of spastic CP, quadriparetic CP (QCP) is the most severe and accounts for 20% of spastic CP cases. Individuals diagnosed with quadriparetic cerebral palsy (QCP) are restricted from participating in daily life activities due to inadequate upper extremity function (spasticity, muscle weakness, inability to perform isolated movements, and limitation of supination movements). In order to correctly evaluate children diagnosed with QCP and determine treatment priorities, it is very important to evaluate them based on the International Classification of Functioning, Disability, and Health (ICF). In the literature, there is no study that evaluates the upper extremity of individuals with isolated QCP based on ICF. The aim of this study is to examine the upper extremity functions of individuals with isolated QCP diagnosis within the framework of ICF.

DETAILED DESCRIPTION:
It is an observational study. Purpose of the study: To examine the upper extremity functions of individuals with an isolated diagnosis of quadriparetic Cerebral Palsy (QCP) within the framework of ICF.

Participants: Children with quadriparetic CP between the ages of 0-17.

Questions:

* What is the relationship between upper extremity spasticity and manual dexterity in children with QCP?
* What is the relationship between manual skills and activities of daily living in children with QCP?

The upper extremities of the patients with QCP will be evaluated within the framework of ICF. Body structure and functions will be evaluated with the Modified Ashworth Scale (MAS), activities with the Manual Ability Classification System (MACS), and participation with the Functional Independence Measure for Children (WeeFIM). The evaluations will be made by physiotherapists experienced in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* The age of the cases is between 0-17,
* They have been diagnosed with quadriparetic CP,
* The participants and parents want to participate in the study voluntarily.

Exclusion Criteria:

* Having different types of CP such as dyskinetic, ataxic and mixed type,
* Having spastic diparetic or hemiparetic type CP,
* Having any history of surgery on the musculoskeletal system,
* Having received Botulinum Toxin injection within the last 6 months.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twenty quadriparetic children with CP, aged 0-17 years, will be included in the study for upper extremity evaluation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | baseline
  It is a 6-point scale that measures the resistance of the muscle to passive movement by passively moving it through the normal range of motion of the joint. Within the scope of the study, the upper extremity muscles; shoulder flexors, shoulder extensors, elbow flexors, elbow extensors, forearm pronators, wrist flexors, wrist extensors, and fingers will be evaluated with MAS.
Manual Ability Classification System (MACS) | baseline
  It is used to classify how children with CP use their hands to handle objects in daily activities. The MACS identifies 5 levels. The MACS levels are functional descriptions based on a child's usual, self-initiated ability to handle objects in daily activities. The levels are based on children's ability to handle objects independently and their need for assistance or adaptations to perform manual activities in daily life.
Functional Independence Measure for Children (WeeFIM) | baseline
  It was developed to assess the functional independence levels of children with developmental disabilities in their daily living activities. The scale consists of 6 sections: self-care (6 items), sphincter control (2 items), transfers (3 items), movement (2 items), communication (2 items), and social and cognitive status (3 items). There are a total of 18 items in the sections. All items in the sections are scored from 1 to 7. 1 point indicates full dependency; 7 points indicate full independence. A total of 18 (full dependency) points and a maximum of 126 (full independence) points can be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Yıldızdağı, Principal Investigator — Acıbadem Atunizade Hospital
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, AA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.